CLINICAL TRIAL: NCT03851302
Title: Effects of Remote Ischemic Conditioning on Hand Use in Individuals With Spinal Cord Injury and Amyotrophic Lateral Sclerosis: A Preliminary Study
Brief Title: Effects of Remote Ischemic Conditioning on Hand Use in Individuals With SCI and ALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bronx VA Medical Center (U.S. Federal Agency)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Noam Y. Harel, Principal Investigator, Bronx VA Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HAR-18-47; R03HD097709 (NIH)
Record Dates: First submitted 2019-02-16; First posted 2019-02-22 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Spinal Cord Injuries; Amyotrophic Lateral Sclerosis
Keywords: Remote ischemic conditioning; Neuroplasticity; transcranial magnetic stimulation
MeSH Terms: conditions — Spinal Cord Injuries; Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Able bodied: Able bodied: sham first, then active (Experimental): Subjects without SCI or ALS. Sham first, then active.
  Interventions: Other: Active Remote Ischemic Conditioning; Other: Sham Remote Ischemic Conditioning; Other: Isometric hand exercise
- Able bodied: active first, then sham (Experimental): Subjects without SCI or ALS. Active first, then sham.
  Interventions: Other: Active Remote Ischemic Conditioning; Other: Sham Remote Ischemic Conditioning; Other: Isometric hand exercise
- Spinal Cord Injured: active first, then sham (Experimental): Participants with Spinal Cord Injury. Active first, then sham.
  Interventions: Other: Active Remote Ischemic Conditioning; Other: Sham Remote Ischemic Conditioning; Other: Isometric hand exercise
- Spinal Cord Injured: sham first, then active (Experimental): Participants with Spinal Cord Injury. Sham first, then active.
  Interventions: Other: Active Remote Ischemic Conditioning; Other: Sham Remote Ischemic Conditioning; Other: Isometric hand exercise
- Amyotrophic lateral sclerosis: active first, then sham. (Experimental): Participants with amyotrophic lateral sclerosis. Active first, then sham.
  Interventions: Other: Active Remote Ischemic Conditioning; Other: Sham Remote Ischemic Conditioning; Other: Isometric hand exercise
- Amyotrophic lateral sclerosis: sham first, then active. (Experimental): Participants with amyotrophic lateral sclerosis. Sham first, then active.
  Interventions: Other: Active Remote Ischemic Conditioning; Other: Sham Remote Ischemic Conditioning; Other: Isometric hand exercise

INTERVENTIONS:
Other: Active Remote Ischemic Conditioning — The active RIC protocol involves 5 cycles of 5-min inflation and 5-min deflation on the non-target arm. The active RIC will be achieved via blood pressure cuff inflation to 200 mmHg.
Other: Sham Remote Ischemic Conditioning — The sham RIC protocol involves 5 cycles of 5-min inflation and 5-min deflation on the non-target arm. The sham RIC will be achieved via blood pressure cuff inflation to 10 mmHg below the subjects' diastolic blood pressure which would not cause the blood occlusion.
Other: Isometric hand exercise — Participants will be instructed to pinch a dynamometer with thumb and index finger at different intensities and durations. The intensities of pinch force will be 10%, 25%, and 50% of the maximal voluntary contraction (MVC). For each intensity, durations of 2, 4, and 6 s will be employed, which resulted in nine different combinations delivered in pseudorandom order. Participants will perform 2 sets of the isometric hand exercise (18 pinches in total). The interval between each pinch will be 2 seconds, with 30 second intervals between each set.

SUMMARY:
Rehabilitation interventions such as physical training and neural stimulation after spinal cord injury (SCI) have been shown to increase neural plasticity. However, both physical training and neural stimulation require a large number of repetitions, and the retention of the intervention effects may be fleeting. In this proposal the investigators will test Remote ischemic conditioning (RIC), which has been shown to promote neural plasticity and has practical and theoretical advantages. RIC consists of transiently restricting blood flow to any 'remote' limb using a blood pressure cuff. This induces several of the body's systemic defensive reactions. RIC has been shown to improve motor learning. The investigators propose that RIC alters motor pathway excitability through a combination of systemic increases in plasticity-promoting factors and inhibition of inflammatory factors. The investigators have designed a clinical trial to test this hypothesis in 8 persons with SCI and 8 able-bodied controls. All participants will receive active/sham RIC plus a hand exercise. The investigators will measure effects on blood pressure, motor neuron excitability, and systemic inflammatory markers before and after RIC as well as after hand exercise. Starting July 2021, we will also enroll 5 individuals with Amyotrophic lateral sclerosis (ALS) in this study.

DETAILED DESCRIPTION:
Most spinal cord injuries (SCI) are not full transections, indicating that there are residual nerve circuits after injury. Rehabilitation interventions after SCI, including physical training and neural stimulation, have been shown to reorganize motor pathways in the brain, corticospinal tract (CST), and at the spinal level; a process called neural plasticity. Functional improvement due to neural plasticity after SCI could be from enhanced excitability of residual neural circuits, or axon sprouting which has been shown in animal studies. However, both physical training and neural stimulation require a large number of repetitions, and the retention of the intervention effects may be fleeting. Therefore, the need remains for an effective approach to synergistically improve neuroplasticity in combination with other interventions. Remote ischemic conditioning (RIC) has been shown to promote neural plasticity and may have practical and theoretical advantages, which include: 1) RIC requires minimal equipment, (a timer and a manual blood pressure device); and 2) RIC has been shown to promote Hypoxia-inducible factor 1a (HIF-1a) and anti-inflammatory mediators which possibly promote neuroplasticity. In fact, One recent study has demonstrated in able-bodied subjects that introducing RIC before a motor learning intervention had a greater and longer-lasting effect on improving motor performance compared to sham conditioning prior to motor learning. In this proposed study, the investigators will investigate RIC coupled with physical training to promote neuroplasticity in hand muscles after cervical SCI. This will be the first study to introduce RIC in SCI population. The investigators hypothesize that RIC will acutely synergize with motor task training via increasing corticospinal excitability. Identifying the underlying mechanisms responsible for increasing corticospinal excitability, such as 1) increased cortical firing, 2) strengthened synaptic transmission, 3) improved spinal motor neuron recruitment or 4) other mechanisms is an important step for promotion of functional recovery after neurological injury. Aim 1: To determine the effects of active versus sham RIC prior to one bout of muscle contraction exercise on motor corticospinal excitability at the abductor pollicis brevis (APB) muscle. The investigators will also assess intra-cortical facilitation/inhibition and peripheral nerve conduction profiles to localize the level of changes in corticospinal excitability. Aim 2: To investigate effects of active versus sham RIC on systemic inflammatory mediators in individuals with SCI. Individuals living with SCI often show signs of chronic inflammation and other aspects of dysregulated immune system function. Studies in able-bodied adults have shown that a single application of RIC can suppress inflammatory gene expression in circulating leukocytes 15 min and 24h later. Upregulation of inflammatory cytokines is associated with decreased expression of genes that promote neuroplasticity, such as brain-derived neurotrophic factor (BDNF). Here, the investigators will determine if RIC decreases systemic inflammation in persons with chronic SCI, as it does in able-bodied individuals, by measuring a subset of inflammatory mediators in the blood pre- and post-RIC. Aim 3: To determine changes in heart rate (HR), blood pressure (BP) and oxygen saturation (SaO2) during active versus sham RIC in individuals with incomplete cervical SCI and able-bodied subjects. RIC has been shown to be safe in the healthy population as well as in individuals with heart disease and even critically ill patients with subarachnoid hemorrhage. However, there are no data describing the safety of RIC in persons with SCI. Damage to the autonomic nervous system (ANS) contributes to cardiovascular dysregulation and may alter physiological responses to RIC. In addition, the SCI population, particularly those with cervical SCI, has widespread sensory impairment, including a limited ability to feel pain/discomfort. The investigators will not only real-time record HR, BP and SaO2 responses during RIC, but also document the pain scale and any adverse effects of RIC in individuals with cervical SCI and able-bodied subjects.

ELIGIBILITY:
Able-bodied participants

1. Age between 18 and 75 years;
2. No known central or peripheral neurological disease or injury.

SCI participants

Inclusion Criteria:

1. Age between 18 and 75 years;
2. Chronic (more than 12 months since injury) motor-incomplete SCI between neurological levels C2-C8
3. Detectable F-wave responses of the left or right abductor pollicis brevis (APB) to median nerve stimulation;
4. Detectable motor evoked potentials in left or right APB muscles to transcranial magnetic stimulation;
5. Able to perform thumb-middle finger opposition pinch task with detectable APB EMG muscle activity.

ALS participants

1. Age between 21 and 75 years;
2. Diagnosis of probable or definite ALS.
3. Incomplete weakness of left or right wrist or hand muscles: score of 2, 3, or 4 (out of 5) on manual muscle testing of finger extension, finger flexion, or finger abduction.
4. Detectable motor evoked potentials in left or right APB muscles to transcranial magnetic stimulation;
5. Able to perform thumb-middle finger opposition pinch task with detectable APB electromyography (EMG) muscle activity.

Exclusion Criteria:

1. Multiple spinal cord lesions;
2. History of seizures;
3. Use of medications that significantly lower seizure threshold, such as amphetamines and bupropion;
4. History of implanted brain/spine/nerve stimulators, aneurysm clips, or cardiac pacemaker/defibrillator;
5. Any extremity soft tissue, orthopedic, or vascular condition or injury that may contraindicate remote limb ischemic conditioning (RLIC) (uncontrolled hypertension, peripheral vascular disease, hematological disease, severe hepatic or renal dysfunction);
6. Any other contraindication to undergoing magnetic resonance imaging (except for claustrophobia);
7. Clinically significant infection of any kind (urinary tract, pulmonary, skin or other)
8. Significant coronary artery or cardiac conduction disease;
9. Open skin lesions over the neck, shoulders, or arms;
10. Pregnancy
11. Unsuitable for study participation as determined by study physician. In addition, a medical record review will be conducted to identify any other medical concerns that might increase the risks associated with participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Kuang Wu, PT, PhD, Principal Investigator — James J. Peters VA Medical Center
Locations (1):
- James J. Peters VA Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
A Limited Dataset (LDS) will be shared in electronic format pursuant to a VA-approved Data Use Agreement. Individually Identifiable Data will be shared pursuant to valid HIPAA Authorization, Informed Consent, and an appropriate written agreement limiting use of the data to the conditions as described in the authorization and consent, and a written assurance from the recipient that the information will be maintained in accordance with the security requirements of 38 Code of Federal Regulations (CFR) Part 1.466.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Available now once above stipulations met.
Access Criteria: Available now once above stipulations met.

REFERENCES:
- [Derived] Wu YK, Harel NY, Wecht JM, Bloom OE. Effects of Remote Ischemic Conditioning on Hand Engagement in individuals with Spinal cord Injury (RICHES): protocol for a pilot crossover study. F1000Res. 2021 Jun 10;10:464. doi: 10.12688/f1000research.52670.2. eCollection 2021. PMID 35342620

RESULTS

PARTICIPANT FLOW:
Groups:
- Able Bodied: Sham First Visit, Active Second Visit: Subjects without spinal cord injury (SCI) or amyotrophic lateral sclerosis (ALS).
  Sham first visit (1 day). Washout (2 weeks). Active second visit (1 day).
- Able Bodied: Active First Visit, Sham Second Visit: Subjects without spinal cord injury (SCI) or amyotrophic lateral sclerosis (ALS).
  Active first visit (1 day). Washout (2 weeks). Sham second visit (1 day).
- Spinal Cord Injury: Active First Visit, Sham Second Visit: Participants with spinal cord injury. Active first visit (1 day). Washout (2 weeks). Sham second visit (1 day).
- Spinal Cord Injury: Sham First Visit, Active Second Visit: Participants with spinal cord injury. Sham first visit (1 day). Washout (2 weeks). Active second visit (1 day).
- Amyotrophic Lateral Sclerosis: Active First Visit, Sham Second Visit: Participants with amyotrophic lateral sclerosis. Active first visit (1 day). Washout (2 weeks). Sham second visit (1 day).
- Amyotrophic Lateral Sclerosis: Sham First Visit, Active Second Visit.: Participants with amyotrophic lateral sclerosis. Sham first visit (1 day). Washout (2 weeks). Active second visit (1 day).
Period: Screening (1 Day)
Arm/Group | Able Bodied: Sham First Visit, Active Second Visit | Able Bodied: Active First Visit, Sham Second Visit | Spinal Cord Injury: Active First Visit, Sham Second Visit | Spinal Cord Injury: Sham First Visit, Active Second Visit | Amyotrophic Lateral Sclerosis: Active First Visit, Sham Second Visit | Amyotrophic Lateral Sclerosis: Sham First Visit, Active Second Visit.
Started | 4 | 5 | 4 | 5 | 3 | 0
Completed | 4 | 5 | 3 | 3 | 3 | 0
Not Completed | 0 | 0 | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Screened out | 0 | 0 | 1 | 1 | 0 | 0
Period: First Intervention (1 Day)
Arm/Group | Able Bodied: Sham First Visit, Active Second Visit | Able Bodied: Active First Visit, Sham Second Visit | Spinal Cord Injury: Active First Visit, Sham Second Visit | Spinal Cord Injury: Sham First Visit, Active Second Visit | Amyotrophic Lateral Sclerosis: Active First Visit, Sham Second Visit | Amyotrophic Lateral Sclerosis: Sham First Visit, Active Second Visit.
Started | 4 | 5 | 3 | 3 | 3 | 0
Completed | 3 | 5 | 3 | 3 | 3 | 0
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Period: Washout (at Least 2 Weeks)
Arm/Group | Able Bodied: Sham First Visit, Active Second Visit | Able Bodied: Active First Visit, Sham Second Visit | Spinal Cord Injury: Active First Visit, Sham Second Visit | Spinal Cord Injury: Sham First Visit, Active Second Visit | Amyotrophic Lateral Sclerosis: Active First Visit, Sham Second Visit | Amyotrophic Lateral Sclerosis: Sham First Visit, Active Second Visit.
Started | 3 | 5 | 3 | 3 | 3 | 0
Completed | 3 | 5 | 3 | 3 | 3 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | Able Bodied: Sham First Visit, Active Second Visit | Able Bodied: Active First Visit, Sham Second Visit | Spinal Cord Injury: Active First Visit, Sham Second Visit | Spinal Cord Injury: Sham First Visit, Active Second Visit | Amyotrophic Lateral Sclerosis: Active First Visit, Sham Second Visit | Amyotrophic Lateral Sclerosis: Sham First Visit, Active Second Visit.
Started | 3 | 5 | 3 | 3 | 3 | 0
Completed | 3 | 5 | 3 | 3 | 3 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: One person in Able-bodied Sham-first group withdrew prior to completion. One person in the SCI-Active-first group screened out. One person in the SCI-Sham-first group screened out. One person in the SCI-Sham-first group withdrew prior to completion.
Groups:
- Total: Total of all reporting groups
Arm/Group | Able Bodied: Sham First Visit, Active Second Visit | Able Bodied: Active First Visit, Sham Second Visit | Spinal Cord Injury: Active First Visit, Sham Second Visit | Spinal Cord Injury: Sham First Visit, Active Second Visit | Amyotrophic Lateral Sclerosis: Active First Visit, Sham Second Visit | Amyotrophic Lateral Sclerosis: Sham First Visit, Active Second Visit | Total
Number analyzed (Participants) | 4 | 5 | 3 | 3 | 3 | 0 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (15.3) | 31.4 (7.8) | 49.3 (22.5) | 44.3 (15.3) | 44.7 (20.8) |  | 43.9 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 0 | 0 | 0 |  | 4
  Male | 2 | 3 | 3 | 3 | 3 |  | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 0 | 1 | 0 | 3
  Not Hispanic or Latino | 4 | 3 | 3 | 3 | 2 | 0 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 0 | 0 | 1 | 0 | 4
  White | 2 | 3 | 3 | 3 | 2 | 0 | 13
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 3 | 3 | 3 |  | 18

OUTCOME MEASURES:

1. Primary Outcome: Percent Change of Electromyographic Responses After Remote Ischemic Conditioning (RIC) Plus Hand Isometric Exercise
Description: Response to electrical and magnetic stimulation will be measured via peak-to-peak amplitude (millivolts) in abductor pollicis brevis muscle.
  Percent change of the electromyographic responses was measured immediately after active/sham RIC plus isometric hand exercise in comparison with baseline measurement. The RIC plus hand exercise duration is 60 minutes.
Time Frame: Outcome measured immediately after completion of RIC plus isometric hand exercise. The RIC plus hand exercise duration is 60 minutes.
Population: One AB participant withdrew during the first study visit. One ALS participant had no valid data during the first study visit and then withdrew.
Measure: Mean (Standard Deviation); unit: change (%) from baseline
Groups:
- Able Bodied-Sham: Sham intervention
- Able Bodied-active: Active intervention
- SCI-Sham: Spinal cord injured-sham intervention
- SCI-Active: Spinal cord injured-active intervention
- ALS-sham: Amyotrophic lateral sclerosis - sham intervention.
- ALS - Active: Amyotrophic lateral sclerosis - active intervention.
Arm/Group | Able Bodied-Sham | Able Bodied-active | SCI-Sham | SCI-Active | ALS-sham | ALS - Active
Number analyzed (Participants) | 8 | 8 | 6 | 6 | 2 | 2
change (%) from baseline | 17.4 (57.6) | 22.2 (46.2) | -19.2 (40.1) | 79.7 (120.4) | -6.1 (10.2) | 111.8 (99.0)

2. Secondary Outcome: Percent Change of Electromyographic Responses After RIC But Before Hand Isometric Exercise
Description: Response to electrical and magnetic stimulation was measured via peak-to-peak amplitude (millivolts) in abductor pollicis brevis muscle.
  Percent change of the electromyographic response was measured immediately after active/sham RIC but before isometric hand exercise in comparison with baseline measurement. The RIC duration is 50 minutes.
Time Frame: Outcome measured immediately after completion of RIC. The RIC duration is 50 minutes.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: change (%) from baseline
Arm/Group | Able Bodied-Sham | Able Bodied-active | SCI-Sham | SCI-Active | ALS-sham | ALS - Active
Number analyzed (Participants) | 8 | 8 | 6 | 6 | 2 | 2
change (%) from baseline | 23.5 (60.1) | 21.6 (89.7) | -14.8 (41.2) | 59.9 (127.2) | 52.3 (56.3) | 200.1 (289.8)

3. Secondary Outcome: Percent Change of Electromyographic Responses 15 Mins After RIC Plus Hand Isometric Exercise
Description: Response to electrical and magnetic stimulation was measured via peak-to-peak amplitude (millivolts) in abductor pollicis brevis muscle.
  Percent change of the electromyographic responses was measured 15 mins after active/sham RIC plus isometric hand exercise in comparison with the measurement immediately after active/sham RIC plus isometric hand exercise. The RIC plus hand exercise duration is 60 minutes. Therefore this is 75 minutes post baseline.
Time Frame: Outcome measured 15 minutes after completion of RIC plus isometric hand exercise. The RIC plus hand exercise duration is 60 minutes. Therefore this is 75 minutes post baseline.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: change (%) from baseline
Arm/Group | Able Bodied-Sham | Able Bodied-active | SCI-Sham | SCI-Active | ALS-sham | ALS - Active
Number analyzed (Participants) | 8 | 8 | 6 | 6 | 2 | 2
change (%) from baseline | 15.2 (78.9) | 35.4 (107.5) | -5.1 (36.5) | 204.9 (291.5) | -46.7 (52.6) | -6.7 (63.3)

4. Secondary Outcome: Blood Pressure
Description: The change in mean arterial pressure will be monitored to ensure the stable hemodynamic responses toward the ischemic stimulation.
Time Frame: Mean arterial pressure at baseline and immediately after intervention on the same day. RIC plus hand exercise duration is 60 minutes.
Population: Pre-post data was not collected for other visits.
Measure: Mean (Standard Deviation); unit: change (mm Hg) from baseline
Arm/Group | Able Bodied-Sham | Able Bodied-active | SCI-Sham | SCI-Active | ALS-sham | ALS - Active
Number analyzed (Participants) | 8 | 8 | 3 | 4 | 2 | 3
change (mm Hg) from baseline | 1.8 (4.4) | 4.4 (4.1) | 8.3 (14.6) | 3.4 (4.9) | -5.2 (5.4) | -3.4 (14.7)

5. Secondary Outcome: Heart Rate
Description: The heart rate will be monitored to ensure the stable hemodynamic responses toward the ischemic stimulation.
Time Frame: Heart rate at baseline and immediately after intervention on the same day. RIC plus hand exercise duration is 60 minutes.
Population: Pre-post data was not collected for other visits.
Measure: Mean (Standard Deviation); unit: change (beats per minute) from baseline
Arm/Group | Able Bodied-Sham | Able Bodied-active | SCI-Sham | SCI-Active | ALS-sham | ALS - Active
Number analyzed (Participants) | 8 | 8 | 2 | 4 | 2 | 3
change (beats per minute) from baseline | -0.8 (5.1) | -4.4 (5.7) | -5.0 (0.7) | 1.5 (10.1) | -6.0 (2.8) | -3.2 (3.8)

6. Secondary Outcome: Oxygen Saturation
Description: The pulse oximetry satuation will be monitored to ensure the stable respiratory responses toward the ischemic stimulation.
Time Frame: Pulse oximetry at baseline and immediately after intervention on the same day. RIC plus hand exercise duration is 60 minutes.
Population: Pre-post data was not collected for other visits.
Measure: Mean (Standard Deviation); unit: change (% saturation) from baseline
Arm/Group | Able Bodied-Sham | Able Bodied-active | SCI-Sham | SCI-Active | ALS-sham | ALS - Active
Number analyzed (Participants) | 7 | 7 | 2 | 4 | 2 | 3
change (% saturation) from baseline | 0.4 (1.4) | 0.6 (1.4) | 1.3 (0.4) | 0.3 (1.3) | 0 (1.4) | 2.3 (2.1)

7. Other Pre Specified Outcome: Inflammatory Mediators: the Intensity of the Gene Expression of Toll-like Receptor (TLR) Signal Pathway.
Description: The blood samples will be collected before and after RIC to analyze on the changes of inflammatory mediators on the intensity of the gene expression related to Toll-like receptor (TLR) signal pathway.
Time Frame: Change in mediator level between baseline measurement and immediately after completion of RIC. RIC duration is 50 minutes.
Reporting Status: Not Posted, anticipated posting 2026-07

ADVERSE EVENTS:
Time Frame: 24 hours
Groups:
- ALS-Active: Amyotrophic lateral sclerosis - sham interven
Arm/Group | Able Bodied-Sham | SCI-Sham | ALS-Sham | Able Bodied-Active | SCI-Active | ALS-Active
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/6 | 0/2 | 0/8 | 0/6 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/6 | 0/2 | 0/8 | 0/6 | 0/3
Other Adverse Events (participants affected / at risk) | 5/9 | 1/6 | 0/2 | 5/8 | 2/6 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Able Bodied-Sham (N=9) | SCI-Sham (N=6) | ALS-Sham (N=2) | Able Bodied-Active (N=8) | SCI-Active (N=6) | ALS-Active (N=3)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Head or scalp pain from transcranial magnetic stimulation
Mood change (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — transient subjective 'spaciness'
Paresthesias (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 1 (1) — Tingling sensations

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-24): https://cdn.clinicaltrials.gov/large-docs/02/NCT03851302/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-16): https://cdn.clinicaltrials.gov/large-docs/02/NCT03851302/ICF_001.pdf